CLINICAL TRIAL: NCT05549349
Title: ANGH Prospective Cohort of Mild and Severe Acute Biliary Pancreatitis
Acronym: CAPABLES
Status: Terminated | Type: Observational
Why Stopped: Studies are finshed
Sponsor: Julia TRAVAGLI (Other)
Responsible Party: Sponsor-Investigator, Julia TRAVAGLI, PhD, Poissy-Saint Germain Hospital
Organization: Poissy-Saint Germain Hospital (Other)
Other Study IDs: 2022-A00303-40
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acute Biliary Pancreatitis
MeSH Terms: interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cholecystectomy during hospitalization: In this group, patients will have their cholecystectomy during the initial hospitalization. We will look at the mode of feeding between the biliary crisis and the cholecystectomy.
  Interventions: Procedure: Cholecystectomy
- Delayed cholecystectomy: In this group, patients will have their cholecystectomy deferred from their initial hospitalization for various reasons. They will be seen again 3 months after leaving hospital. They will or will not have been cholecystectomized during this interval. Their mode of feeding as well as biliary events will be studied.
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Gallbladder removal

SUMMARY:
The main objective of this work is to evaluate the recurrence of biliary episodes before cholecystectomy (hepatic colic, lithiasic migration, cholangitis, cholecystitis, pancreatitis, necrosis infections) in patients with acute biliary pancreatitis of any severity depending on the type of nutrition (oral, enteral or parenteral).

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is one of the frequent causes of hospitalization in gastroenterology with an annual incidence of 13-45 cases per 100,000 patients. If we refer to the data in the white paper, hospitalizations for abdominal emergencies, such as PA, take place in at least 60% of cases in General Hospital Centers (CHG). Among these AP, approximately 40% of AP are secondary to a biliary lithiasis pathology. The main modalities of the initial management of AP have been the subject of several national and international recommendations and consensuses. Although it is well accepted that early refeeding during the first 48 hours reduces the appearance of a systemic inflammatory response syndrome (SIRS) or a collection infection, the feeding methods in the event of pancreatitis Acute biliary (ABP) during the acute phase using the oral route if it is tolerated or the enteral route by nasogastric tube before cholecystectomy remains debated.

Thus, in case of delayed cholecystectomy after AP, there is no consensus on the feeding methods after the acute phase (oral or enteral) until cholecystectomy nor on the benefit of a prophylactic endoscopic sphincterotomy in the absence of cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years old
* Affiliated to a social security scheme.
* Patients with acute biliary pancreatitis

Exclusion Criteria:

* Patients with chronic pancreatitis
* Patients with a previous cholecystectomy
* Patients under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of patients will be done in the gastroenterology departments of participating Hospitals. Information to patients will be provided by an investigator from the service.
  Participation in this study will be offered to all patients fulfilling the inclusion and non-inclusion criteria. A specific written information note as well as clear and honest oral information will be given to patients meeting the inclusion criteria, before collecting their non-objection.
  After collection of the patient's non-objection and allocation of a patient code, the investigator or his representative will complete an observation book (Case Report Form in English, CRF). This observation book will include clinical and paraclinical data from the patient's medical file.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
biliary events | 3 month
  Assess the recurrence of biliary events before cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Frederick MORRYOUSSEF, MD, Principal Investigator — Poissy
Locations (1):
- MORRYOUSSEF Frederick, Poissy, France

IPD SHARING:
Plan to Share IPD: Undecided